CLINICAL TRIAL: NCT05685550
Title: Safety and Efficacy Analysis of Oral Etoposide Combined With Anlotinib and Envafolimab in First-line Treatment of Elderly Patients With Small Cell Lung Cancer/ Open-label, Single-arm, Exploratory Phase II Clinical Study
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS-2022-0048
Record Dates: First submitted 2023-01-03; First posted 2023-01-17 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Progression Free Survival(PFS)
MeSH Terms: interventions — anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Etoposide capsules in combination with Anlotinib and Envafolimab
  Interventions: Drug: Toposide capsules combined with Anlotinib and Envafolimab group

INTERVENTIONS:
Drug: Toposide capsules combined with Anlotinib and Envafolimab group — Elderly patients with extensive SCLC were given etoposide capsules 100mg PO qd*7d and Envafolimab 300mg/ time IH Q3W in combination with Anlotinib 12mg PO qd*14d. Based on the safety and other data from the subjects, the combination regimen was administered for 4 to 6 cycles, with a maximum of 6 cycles. In principle, at least 4 cycles were required unless chemotherapy-related toxicity necessitated early termination. Subsequently, patients without evidence of disease progression received maintenance therapy with Envafolimab plus Anlotinib until disease progression, intolerable adverse events, or death.
  Other Names: Combined treatment group

SUMMARY:
This study aims to explore the safety and efficacy of etoposide capsules combined with Anlotinib and Envafolimab in elderly patients with extensive small cell lung cancer.This is a single-center, single-arm exploratory clinical study. 30 patients with extensive small-cell lung cancer are scheduled to be enrolled. Treatment regimen is etoposide capsule 100mg PO qd*7d, Anlotinib 12mg PO qd*14d, Envafolimab 300mg/ IH Q3W. Based on the safety and other data from the subjects, the combination regimen was administered for 4 to 6 cycles, with a maximum of 6 cycles. In principle, at least 4 cycles were required unless chemotherapy-related toxicity necessitated early termination. Subsequently, patients without evidence of disease progression received maintenance therapy with envolumab plus anlotinib until disease progression, intolerable adverse events, or death.

DETAILED DESCRIPTION:
The primary objective of this study was to explore the safety and median PFS of etoposide capsules combined with Anlotinib and Envafolimab as first-line treatment in elderly patients with extensive small-cell lung cancer (as assessed by the investigators according to RECIST 1.1 criteria).The secondary objective of this study was to evaluate the OS, ORR, and QOL of etoposide capsules combined with Envafolimab and Anlotinib as first-line treatment in elderly patients with extensive small-cell lung cancer.Exploratory aims are to explore predictive or prognostic biomarkers (tissue and/or plasma) associated with therapeutic response or resistance to disease; Analysis of potential biomarkers in biopsy tissue samples and blood samples after disease progression to explore possible mechanisms of therapeutic resistance. To provide a better treatment plan for elderly patients with extensive small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* 4.1.1. Patients with extensive small cell lung cancer confirmed histologically or cytologically;

4.1.2. Has not received systemic antitumor therapy for small cell lung cancer. If the subject receives adjuvant therapy after completing radical therapy for early small cell lung cancer and the subject relapses the disease, ensure that the interval between the end of adjuvant therapy and the first administration of the study is more than 6 months, and that all toxic reactions caused by adjuvant therapy have recovered (Class 1 according to CTCAE v4.0 criteria, except hair loss).

4.1.3. Male or female ≥65 years old and signed informed consent;

4.1.4. The ECOG performance status ≤3, and the expected survival is greater than 6 months;

4.1.5. There must be at least one measurable target lesion (according to RECIST 1.1).

4.1.6. Good organ function: Laboratory tests meet the following requirements: neutrophil absolute value (ANC) ≥1.5×10^9/L, platelet count ≥100×10^9/L, hemoglobin ≥90 g/L, white blood cell ≥3.0×10^9/L; Liver function: total bilirubin < 1.5 times the upper limit of normal value, AST/SGOT, ALT/SGPT and alkaline phosphatase (ALP) < 2.5 times the upper limit of normal value; If liver metastasis occurs, AST and ALT≤5.0 times the upper limit of normal value; For liver and/or bone metastases, ALP≤5.0 times the upper limit of normal. Renal function: serum creatinine (Scr) ≤1.5 times the upper limit of normal; Urine protein < 2 (+) was detected by routine urine test. If urine protein ≥2 (+) at baseline, 24-hour urine protein quantity must be ≤1.0 g; Coagulation function: International standardized ratio (INR) ≤1.5, and activated partial thromboplastin time (APTT) ≤1.5 times the upper limit of normal value;

4.1.7. Cardiac function: left ventricular ejection fraction (LVEF) ≥50%;

4.1.8 Be able to communicate well with the investigator and follow the study requirements for visits, treatment, laboratory tests and other relevant regulations.

Exclusion Criteria:

* 4.2.1. Previous anti-PD-1, anti-PD-L1, anti-PD-L2, TIGIT or any other antibody or drug therapy specifically targeting T-cell costimulation or checkpoint pathways;

4.2.2. With active pinimeningeal disease or poorly controlled and untreated brain metastases:

Note: Patients with a history of central nervous system metastasis and stable at screening are eligible for admission only if they meet all of the following criteria:

1. Brain imaging at screening showed no evidence of progression, clinically stable for at least 2 weeks, and no evidence of new brain metastases;
2. Has a measurable and/or evaluable disease outside the central nervous system;
3. Corticosteroids are not currently required to treat central nervous system diseases; Steroid discontinuation 3 days prior to initial study treatment; Stable doses of anticonvulsants are permitted;
4. No stereotactic radiation or whole brain radiotherapy was performed within 14 days prior to the first study treatment;

4.2.3. Patients with active autoimmune disease or a history of autoimmune disease that may recur;

Note: Patients with the following diseases are not excluded for further screening:

1. Well-controlled type 1 diabetes mellitus;
2. Hypothyroidism (if controlled with hormone replacement therapy alone);
3. Well-controlled celiac disease;
4. Skin diseases that do not require systemic treatment (e.g. vitiligo, psoriasis, alopecia);
5. Any other disease that is not expected to recur in the absence of an external trigger;

4.2.4. There were any active malignancies within 2 years prior to the first administration of the study drug, except for the specific cancers being studied in this study and locally recurring cancers that have been cured (e.g. resected basal cell or squamous cell skin cancer, superficial bladder cancer, breast cancer in situ).

4.2.5. Any condition requiring systemic corticosteroid therapy (doses greater than 10 mg/ day of prednisone or equivalent) or other immunosuppressant treatment within 14 days prior to the first administration of the study drug.

Note: Patients who are currently using or have previously used any of the following steroid regimens may be enrolled:

1. Adrenalin substitute steroid (prednisone ≤10mg/d or equivalent dose of similar drugs);
2. Minimal systemic uptake of local, ocular, intra-articular, intranasal, and inhaled corticosteroids. c. Short-term (≤7 days) use of corticosteroids for prevention (e.g., allergy to contrast media) or treatment of non-autoimmune conditions (e.g., delayed hypersensitivity caused by contact allergens).

4.2.6. The presence of poorly controlled diabetes mellitus, abnormal laboratory results of potassium, sodium, or corrected calcium > grade 1, or ≥ grade 3 hypoalbuminemia in the 14 days preceding and including the first administration of the study drug.

4.2.7. Poorly controlled pleural effusion, pericardial effusion, or ascites requiring frequent drainage (2 weeks after intervention Internal recurrence).

4.2.8. The presence of interstitial lung disease, non-infectious pneumonia or poorly controlled lung diseases (including pulmonary fibrosis, Acute lung disease) history. Patients with significantly impaired lung function or who require oxygen at baseline must be evaluated for lung function at screening.

4.2.9. Had an infection (including tuberculosis, etc.) requiring systemic antibacterial, antifungal or antiviral treatment within 14 days prior to the first administration of the study drug.

Note: Patients with chronic hepatitis B virus (HBV) or hepatitis C virus (HCV) infection are allowed to receive antiviral therapy.

4.2.10. Chronic HBV carriers with untreated chronic hepatitis B or HBV DNA> 500 IU/mL (> 2500 copies /mL) were present at screening.

Note: Non-active hepatitis B surface antigen (HBsAg) carriers, treated and stable hepatitis B patients (HBV DNA < 500 IU/mL or < 2500 copies /mL) could be enrolled. Patients who are HBsAg positive or have detectable HBV DNA should be managed according to treatment guidelines. Patients who were receiving antiviral therapy at the time of screening should be treated for > 2 weeks prior to enrolling.

4.2.11. Patients with active hepatitis C.

Note: Patients who tested negative for HCV antibodies at screening or who tested positive for HCV antibodies at screening but subsequently tested negative for HCV RNA were enrolled. HCV RNA testing will only be performed in patients who test positive for HCV antibodies. Patients who were receiving antiviral therapy at the time of screening should be treated for > 2 weeks prior to enrolling.

4.2.12. Known history of HIV infection.

4.2.13. Any major surgical procedures were performed within 28 days prior to the first administration of the study drug. Patients must have fully recovered from the toxicity and/or complications of the intervention prior to initial administration of the investigational drug.

4.2.14. Previous allogeneic stem cell transplantation or organ transplantation.

4.2.15. Have any of the following cardiovascular risk factors:

1. Cardiogenic chest pain, defined as moderate pain with limited instrumental activities of daily living, occurred within 28 days (including 28 days) before the first administration of the drug;
2. Occurrence of pulmonary embolism within 28 days (including 28 days) prior to the first administration of the study drug;
3. The study had acute myocardial infarction within 6 months (including 6 months) before the first administration of the drug;
4. A history of New York Heart Association (NYHA) Class III or IV heart failure within 6 months including 6 months prior to initial administration of the drug;
5. Study the occurrence of grade 2 or greater ventricular arrhythmias within 6 months (including 6 months) prior to initial drug administration;
6. Cerebrovascular accidents occurred within 6 months (including 6 months) before the first administration of the study drug;
7. Study the presence of poorly controlled hypertension treated with standard antihypertensive drugs within 28 days (including 28 days) prior to initial drug administration;
8. Study any syncope or seizures within 28 days (including 28 days) prior to initial administration of the drug;

4.2.16. History of severe hypersensitivity to other monoclonal antibodies.

4.2.17. Patients who have previously received systemic therapy (prior adjuvant or neoadjuvant therapy is allowed) or have received any immunotherapy (e.g., interleukin, interferon, thymosin, etc.) or any experimental therapy within 14 days or 5 half-lives prior to the first administration of the study drug, whichever is the older. Or received palliative radiotherapy or other local treatment within 14 days before the study drug was first administered.

4.2.18. Toxicity from previous antitumor therapy has not returned to baseline or stabilized (except for adverse events unlikely to pose a safety risk, such as hair loss, neuropathy or abnormal results of specific laboratory tests).

4.2.19. Live vaccine was administered within 28 days (including 28 days) prior to the first administration of the study drug.

Note: Seasonal influenza vaccines are usually inactivated and are permitted for use. The vaccine used in the nasal cavity is a live vaccine and should not be used.

4.2.20. There are underlying medical conditions (including abnormal laboratory results), alcohol or drug abuse or dependence that adversely affect study drug administration, or affect the interpretation of drug toxicity or AE, or lead to inadequate compliance with study execution.

4.2.21. Pregnant or lactating women.

4.2.22. Also participate in another therapeutic clinical trial.

Note: Participation in both observational and non-interventional studies is permitted. In addition, patients who have completed drug therapy in clinical studies and are in the follow-up period are eligible for this study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
PFS (Progression-Free-Survival) | 30 months
  The time from randomization to tumor progression or death.The efficacy of this study was determined according to Recist version 1.1 criteria.

SECONDARY OUTCOMES:
OS (Overall survival time) | 30 months
  The time of death from all causes for all patients from the date of randomization.The efficacy of this study was determined according to Recist version 1.1 criteria.
ORR (Objective response rate) | 30 months
  Defined as complete response and partial response (CR+PR).The efficacy of this study was determined according to Recist version 1.1 criteria.
QOL (Quality of Life) assessed by the QLQ-C30 scale | 30 months
  It mainly refers to the state assessment of individual physiological, psychological and social functions, namely, health quality. The quality of life was assessed by the QLQ-C30 scale
The Adverse Events | 30 months
  AEs are any adverse medical events that occur in a subject or clinical subject and is not necessarily causally related to the treatment. Safety assessment in this study was conducted by the investigator in accordance with the definition of NCI-CTC version 3.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Cancer Hospital Airport Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No